CLINICAL TRIAL: NCT07116772
Title: A Prospective Longitudinal Study of Growth, Development, Fertility and Reproductive Outcomes Among Adolescents and Young Adults With Sickle Cell Anemia With Hydroxyurea
Brief Title: Serial Assessment of Fertility Experiences
Acronym: SAFE
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Caribbean Institute for Health Research, University of West Indies (Unknown); Centro de Obstetricia y Ginecologia Recruiting Santo Domingo, Dominican Republic (Unknown)
Responsible Party: Sponsor
Other Study IDs: SAFE
Record Dates: First submitted 2025-07-23; First posted 2025-08-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Anemia
Keywords: Hydroxyurea; Fertility; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and FTA dried blood spots.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell Anemia: Those with sickle cell anemia (SCA).

SUMMARY:
The SAFE study is a long-term research project that watches people with sickle cell anemia (SCA) over time. The main goal is to see how a medicine called hydroxyurea affects their growth, puberty, and ability to have children. A second goal is to see how hydroxyurea affects pregnancy outcomes, by comparing people who take the medicine to those who don't.

DETAILED DESCRIPTION:
Hydroxyurea is a medicine that helps people with sickle cell anemia (SCA), a serious blood disease. It works by increasing a special type of hemoglobin (called fetal hemoglobin) that helps prevent sickle cell problems.

This medicine is especially helpful in places where it's hard to get safe blood transfusions. Studies from around the world have shown that hydroxyurea is safe and can reduce serious health problems caused by SCA (like pain, strokes, and lung issues). It can also help people with SCA live longer, healthier lives.

However, the investigators still don't know everything about how hydroxyurea affects long-term growth, puberty, fertility, or pregnancy; especially in areas with fewer medical resources.

To learn more, researchers are planning a large international study. They will follow people with SCA over time to see how hydroxyurea affects their development, ability to have children, and pregnancy outcomes. Participants will visit the clinic every few months for check-ups, blood tests, and other health assessments. Girls who have started their periods will take pregnancy tests every six months, and boys may be asked to provide a semen sample if they agree. Everyone will also answer questions about their health and fertility regularly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented sickle cell anemia (SCA).
* At least 8 years of age at the time of enrollment.
* Enrolled on the EXTEND or SACRED study.
* Provide informed consent.
* Able to take part in all parts of the study, including treatments, check-ups, and follow-up visits.

Exclusion Criteria:

* Currently taking part in another treatment study (not EXTEND or SACRED).
* Has received other treatments for sickle cell disease in the past 6 months.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with sickle cell anemia who are at least 8 years old and seen in Jamaica and Dominican Republic.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2035-05-19 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes | From enrollment up to 10 years after enrollment.
  The number of people who experience serious health events like pregnancy, stroke, cancer, or death.

SECONDARY OUTCOMES:
Female Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Female fertility potential will be measured using serum anti-mullerian hormone (physiologic parameter)
Female Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Female ability to conceive will be assessed using incidence of pregnancy (questionnaire)
Female Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Outcomes of pregnancy will be categorized as either abortion or live birth (questionnaire)
Female Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Mode of delivery will be categorized as vaginal or c-section (questionnaire)
Female Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Prematurity of infant will be categorized as premature or full term (questionnaire)
Female Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Weight of infant will be categorized as normal birth weight or low birth weight (questionnaire)
Male Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Male fertility potential will be measured using sperm analysis (physiologic parameter)
Male Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Male ability to conceive will be assessed using incidence of impregnated partner (questionnaire)
Male Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Outcomes of pregnancy will be categorized as either abortion or live birth (questionnaire)
Male Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Mode of delivery will be categorized as vaginal or c-section (questionnaire)
Male Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Prematurity of infant will be categorized as premature or full term (questionnaire)
Male Reproductive Potential and Outcomes | From enrollment up to 10 years after enrollment.
  Weight of infant will be categorized as normal birth weight or low birth weight (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Russell E Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- Centro de Obstetricia y Ginecologia, Santo Domingo, Dominican Republic
- Caribbean Institute for Health Research, University of West Indies, Kingston, Jamaica
- Buganda Medical Centre, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: No
Study data will be collected and managed using REDCap™ electronic data capture tools. REDCap™ is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. The REDCap™ system is available for use through institutions participating in the REDCap™ consortium. Cincinnati Children's Hospital Medical Center serves as the home institution to allow the REDCap™ system for de-identified data collection in the SAFE study.

REFERENCES:
- See also: SACRED ClinicalTrials.gov Posting — https://clinicaltrials.gov/study/NCT02769845?cond=Sickle%20Cell%20Anemia&term=SACRED&rank=1
- See also: EXTEND ClinicalTrials.gov Posting — https://clinicaltrials.gov/study/NCT02556099?cond=Sickle%20Cell%20Disease&term=EXTEND&rank=1